CLINICAL TRIAL: NCT04805463
Title: Evaluation of the Effects of PRF, CGF and AFG Application on Wound Healing Following Gingivectomy and Gingivoplasty Operations: a Randomized Controlled Clinical Trial
Brief Title: Different Platelet Concentrates After Gingivectomy and Gingivoplasty Evaluation of Its Effect on Early Wound Healing.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Esra Bozkurt, RA, Inonu University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2019/216
Record Dates: First submitted 2021-03-16; First posted 2021-03-18 (Actual); Last update posted 2021-03-23 (Actual); Status verified 2021-03

CONDITIONS: Wound Heal; Gingival Overgrowth; Gingival Enlargement; Platelet Rich Fibrin
Keywords: Autologous fibrin glue; Concentrated growth factor; Gingivectomy; Gingivoplasty; Platelet rich fibrin
MeSH Terms: conditions — Gingival Overgrowth; Gingival Hyperplasia | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Split mouth design was used in the study. The chin was divided into lower, upper and right, and left anterior regions. The distribution of the platelet concentrate and control group to be used after gingivectomy and gingivoplasty was randomly decided.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- control group (Experimental): After gingivectomy and released into the secondary wound healing gingivoplasty group.
  Interventions: Other: Control group
- PRF group (Experimental): The group in which PRF was applied to the wound surface after gingivectomy and gingivoplasty.
  Interventions: Other: PRF group
- CGF group (Experimental): The group in which CGF was applied to the wound surface after gingivectomy and gingivoplasty.
  Interventions: Other: CGF group
- AFG group (Experimental): The group in which AFG was applied to the wound surface after gingivectomy and gingivoplasty.
  Interventions: Other: AFG group

INTERVENTIONS:
Other: Control group — The group that did not undergo any procedure after gingivectomy and gingivoplasty operation. Periodontal pack (Coe-Pak, GC America Inc, IL, USA) was applied to the wound area.
  Arms: control group
Other: PRF group — The group in which PRF is applied to the wound area after gingivectomy and gingivoplasty operation. Periodontal pack (Coe-Pak, GC America Inc, IL, USA)was applied over the PRF.
  Arms: PRF group
Other: CGF group — The group in which CGF is applied to the wound area after gingivectomy and gingivoplasty operation. Periodontal pack (Coe-Pak, GC America Inc, IL, USA) was applied over the CGF.
  Arms: CGF group
Other: AFG group — The group in which AFG is applied to the wound area after gingivectomy and gingivoplasty operation. Periodontal pack (Coe-Pak, GC America Inc, IL, USA) was applied over the AFG.
  Arms: AFG group

SUMMARY:
The aim of this study was to evaluate the effect of PRF, CGF and AFG application on early wound healing after gingivectomy and gingivoplasty operations. In the study designed split mouth, gingivectomy and gingivoplasty surgery were performed on 19 patients. The postoperative PRF, CGF, and AFG applied areas were compared with the control regions. 0th,7 th,14 th and 28 th on the days, the surgical area was painted with mira-2-tone solution and evaluated in the ImageJ program. Measurements of clinical periodontal parameters including PI, GI, SC and SD were recorded at the beginning, after IPT and 28 days after the operation. Wound healing was evaluated with H2O2 test, VAS-Pain, and LTH index on 7th, 14th and 28th days. The patients were asked to evaluate their aesthetic perceptions on the VAS aesthetic scale.

DETAILED DESCRIPTION:
Study design and patient selection

In this randomized, controlled, split-mouth (lower, upper jaw, right and left anterior regions) clinical study, who applied to İnönü University Faculty of Dentistry Department of Periodontology between January 2020 and May 2020, due to gingival problems, chronic examination was performed. included individuals diagnosed with inflammatory gingival enlargement.

All patients received initial periodontal therapy (BPT). The patients were called for control after 2 weeks and surgery was planned for the patients who provided adequate oral hygiene. In our study, the vertical DM index, first described by Goaz and Angelopoulos, and later modified by Damm and Miller (DM), was used to classify the gingival enlargement in the vertical direction (1). In order to classify the bucco-lingual gingival growths in the interdental papillae, the horizontal MB index, first described by Seymour et al. And later modified by Miranda and Brunet (MB), was used (2). As a result of the measurements made, grades other than score 0 according to the DB and MB indices were accepted as having gingival enlargement. The distribution of control (n = 19) and three test groups (n = 19, n = 19, n = 19) after gingivectomy and gingivoplasty was randomized (block randomization).

Clinical Measurements

In clinical periodontal evaluation, plaque index (PI) (3), gingival index (GI) (4), bleeding on probing (SC) and probing depth (SD ) measurements were performed at baseline (T0), after BPT (T1) and on the 28th day (T2) after gingivectomy and gingivoplasty operation. Measurements were made in a total of 6 regions of all teeth: mesio-buccal, mid-buccal, disto-buccal, disto-lingual / palatinal, mid-lingual / palatinal and mesio-lingual / palatinal. Clinical periodontal measurements of all teeth of the individuals included in the study were performed by a single investigator (E.B.).

Gingivectomy and gingivoplasty

Before surgery, all patients were gargled with 0.12% chlorhexidine for 1 minute. The incision lines were determined by applying infiltrative anesthesia (Maxicaine Fort) to the areas to be operated, and the external bevel incision was performed with a # 15 scalpel (Broche® Medical scalpel tip; carbon steel) and a Kirkland blade (Hu-Friedy, Chicago, IL, USA). Orban blade (Hu-Friedy, Chicago, IL, USA) was used in the interproximal areas. After the incision was completed, the remaining gum pieces were removed with the help of periodontal curette and microsurgical scissors (Hu-Friedy, Chicago, IL, USA). Then gingivoplasty was performed. After gingivectomy and gingivoplasty, the control areas were left to recover spontaneously. PRF, CGF and AFG were applied to the test areas. Surgical areas in control and test areas were covered with a periodontal pat (Coe-Pak, lsip, IL, USA).

Preparation of platelet-rich fibrin membrane

Blood taken from the antecubital veins of the patients was collected into 10 ml sterile glass-covered plastic tubes (Vacuette serum tubes, Greiner Bio-one) that did not contain anticoagulants. The collected venous blood was placed in the PC-02 (Process, Nice, France) centrifuge device and centrifuged at 3000 rpm for 10 (400xg) minutes (5). The obtained PRF was taken out of the tube, placed in the PRF-BOX and turned into a membrane by compressing with light pressure for about 1 minute. The prepared PRF membranes were applied to the surgical operation area and the operation area was closed with a periodontal pat.

Preparation of concentrated growth factor membrane

Blood taken from the antecubital veins of the patients was collected into 10 ml sterile glass-covered plastic tubes (Vacuette serum tubes, Greiner Bio-one) that did not contain anticoagulants. These tubes were then centrifuged in a centrifuge device (Medifuge; Silfradent srl, Sofia, Italy) using a program with the following features: acceleration for 30 seconds followed by 2 minutes (692xg) at 2700 rpm, 4 minutes (547xg) at 2400 rpm, 2700 rpm. Centrifugation for 4 minutes (592xg) at 3000 rpm for 3 minutes (855xg) and finally deceleration for 36 seconds (6). After centrifugation, CGF was taken from the middle part of the tube, placed in PRF-BOX and turned into a membrane by compressing with light pressure for about 1 minute. Prepared CGF membranes were applied to the surgical operation area and the operation area was closed with a periodontal pat.

Preparation of autologous fibrin glue

Venous blood taken from the patient was transferred to a 9 ml glass-covered plastic tube (Vacuette serum tubes, Greiner Bio-one) that did not contain any anticoagulants. Sohn et al. In the protocol he recommended (7), the venous blood collected in the tube was centrifuged in a centrifuge device (Medifuge, Silfradent, Italy) at 2700 rpm (approximately 692 g) for 2 min. AFG obtained from the upper part of the tube after centrifugation was collected with the help of an injector and transferred to the metal body. The polymerization was allowed for 15-20 minutes. After polymerization was completed, AFG was applied to the surgical operation area and the operation area was covered with a periodontal pat.

Post Operative Care and Suggestion

Patients were advised to protect the wound area with periodontal pats from trauma, not to consume too hot and too cold foods, and to eat soft foods. It was stated that the pat should be kept in the mouth for 1 week, and if the pat was damaged during this period, they should apply to our clinic immediately. Patients were prescribed paracetamol-containing analgesic (Parol 500 mg) and a mouthwash containing 0.12% chlorhexidine to use three times a day for a week. The patients were only advised not to brush their teeth in the operation area for 1 week. It was stated that he should provide oral hygiene in areas that were not operated. They were advised to use an extra soft toothbrush in the area after the pat was removed.

Surface area determination

Mira-2-tone, a plaque staining agent (GMBH & Co., Duisburg, Germany), was used to detect wound surface epithelization at baseline, postoperative 7, 14, and 28 days. Standardized photographs were taken from each patient to evaluate the dark stained areas after staining with Mira-2-tone in the gingiva where epithelialization was not completed and wound healing continued. During the photo shoot, the patients were seated upright and facing straight ahead. All photos were taken by a single person on the same camera (Nikon Coolpix 4500, Tokyo, Japan), at the same distance (20 cm) and light values (ISO-800). The photo size was scaled by using a 10 mm Williams periodontal probe during the photo taking. Wound surface epithelization was calculated using Image J software program (National Institutes of Health, USA ImageJ 1.48V) from the photographs obtained. Each measurement step was done by the same researcher (E.B.) each time. The calibration of the person who made the measurements was performed by repeating the wound surface epithelialization area measurement at one-week intervals on the photo images of 10 patients who had undergone gingivectomy and gingivoplasty surgery and were not included in the study. In these two separate evaluations, the calculations were 95% compatible.

Epithelialization test

In order to evaluate the wound surface epithelization during the healing process, 3% H2O2 was applied to the surface of the operation area with the help of an injector. As a result of the decomposition of H2O2 into water and oxygen through the catalase enzyme released by the blood cells present in the wound area, it was evaluated as "epithelization incomplete" if foaming was observed with oxygen formation, and "epithelization completed" if foaming was not observed . H2O2 test was performed at the controls on the 7th, 14th and 28th days after the operation.

Healing index Landry, Turnbull, and Howley (LTH) index, which classified the healing process according to wound surface redness, presence of bleeding, granulation tissue, epithelization, and suppuration (8). The wound healing process with LTH index was performed at the postoperative 7th, 14th and 28th days.

Postoperative pain and aesthetic

VAS was used for postoperative pain and aesthetic evaluation (9). The patient's 7th, 14th He was asked to evaluate the level of pain he felt from 1 to 10 according to the VAS-Pain (1: low pain, 10: severe pain) scale in the control sessions on the 28th and 28th days. In the control session on the 28th day, the patients were asked to evaluate their aesthetic perceptions from 1 to 10 according to the VAS-Aesthetics (1: dissatisfied, 10: very satisfied) scale.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are systemically healthy, have chronic inflammatory gingival enlargement in the maxillary and mandibular anterior region, and who do not have attachments and bone loss in clinical and radiographic evaluation.

Exclusion Criteria:

* Patients with a history of periodontal treatment in the last 6 months, smokers, those using drugs that may cause gingival enlargement, and pregnant or breastfeeding women were excluded.

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-05-30 (Actual)

PRIMARY OUTCOMES:
Determination of non-epithelialized areas on the wound surface | Postoperative 0, 7, 14 and 28 days, the change of the stained area with the mira-2 tone in the wound surface area was recorded.
  Mira-2 tone solution was used to identify non-epithelialized areas on wound surfaces after gingivectomy and gingivoplasty. Mira-2 tone was applied to the wound surfaces and dark dyed areas were calculated as mm2 in Image j program.
Epithelialization test | The change in wound surface epithelization was evaluated on the 7th, 14th and 28th days postoperatively.
  H2O2 was used to identify non-epithelialized areas. If bubbling is observed after the application of H202 to the wound surface, epithelialization was incomplete, if bubbling was not observed, epithelialization was recorded as completed.
Healing index | Wound healing evaluation with LTH index was performed at the postoperative 7th, 14th and 28th day controls.
  Landry, Turnbull, Howley (LTH) index, which classified the healing process according to wound surface redness, presence of bleeding, granulation tissue, epithelization, and suppuration, was evaluated.
Postoperative pain | Evaluation of VAS-Pain change on postoperative 7th, 14th and 28th days.
  VAS was used for postoperative pain assessment. The patients were asked to evaluate the level of pain from 1 to 10 according to the VAS-Pain (1: low pain, 10: severe pain) scale during the control sessions.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Periodontology, Faculty of Dentistry, Inonu University, Malatya, Battalgazi, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
We have other studies using this data.

REFERENCES:
- [Background] Miranda J, Brunet L, Roset P, Berini L, Farre M, Mendieta C. Prevalence and risk of gingival enlargement in patients treated with nifedipine. J Periodontol. 2001 May;72(5):605-11. doi: 10.1902/jop.2001.72.5.605. PMID 11394395
- [Background] SILNESS J, LOE H. PERIODONTAL DISEASE IN PREGNANCY. II. CORRELATION BETWEEN ORAL HYGIENE AND PERIODONTAL CONDTION. Acta Odontol Scand. 1964 Feb;22:121-35. doi: 10.3109/00016356408993968. No abstract available. PMID 14158464
- [Background] LOE H, SILNESS J. PERIODONTAL DISEASE IN PREGNANCY. I. PREVALENCE AND SEVERITY. Acta Odontol Scand. 1963 Dec;21:533-51. doi: 10.3109/00016356309011240. No abstract available. PMID 14121956
- [Background] Dohan DM, Choukroun J, Diss A, Dohan SL, Dohan AJ, Mouhyi J, Gogly B. Platelet-rich fibrin (PRF): a second-generation platelet concentrate. Part II: platelet-related biologic features. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2006 Mar;101(3):e45-50. doi: 10.1016/j.tripleo.2005.07.009. Epub 2006 Jan 10. PMID 16504850
- [Background] Rodella LF, Favero G, Boninsegna R, Buffoli B, Labanca M, Scari G, Sacco L, Batani T, Rezzani R. Growth factors, CD34 positive cells, and fibrin network analysis in concentrated growth factors fraction. Microsc Res Tech. 2011 Aug;74(8):772-7. doi: 10.1002/jemt.20968. PMID 21780251
- [Background] Sohn D-S, Huang B, Kim J, Park WE, Park CC. Utilization of autologous concentrated growth factors (CGF) enriched bone graft matrix (Sticky bone) and CGF-enriched fibrin membrane in Implant Dentistry. J Implant Adv Clin Dent. 2015;7:11-29.
- [Background] Landry RG. Effectiveness of Benzydamine HC1 in the Treatment of Periodontal Post-surgical Patients: Faculty of Dentistry, University of Toronto; 1985.
- [Background] Crichton N. Visual analogue scale (VAS). J Clin Nurs. 2001;10(5):706-6
- [Result] Miller CS, Damm DD. Incidence of verapamil-induced gingival hyperplasia in a dental population. J Periodontol. 1992 May;63(5):453-6. doi: 10.1902/jop.1992.63.5.453. PMID 1527689